CLINICAL TRIAL: NCT04082949
Title: Evaluation of Clinical Effects of Autologous Fibrin Glue Application as an Adjunct to Nonsurgical Periodontal Treatment of Chronic Periodontitis
Brief Title: Autologous Fibrin Glue Application as an Adjunct to Nonsurgical Periodontal Treatment of Chronic Periodontitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, mustafa özay uslu, Assistant professor, Faculty of Dentistry, Department of Periodontology, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018/45
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Chronic Periodontitis; Periodontal Pocket; Periodontal Attachment Loss; Periodontal Diseases
Keywords: Chronic Periodontitis; Autologous fibrin tissue adhesive; Blood Platelets; Non-surgical periodontal therapy
MeSH Terms: conditions — Chronic Periodontitis; Periodontal Pocket; Periodontal Attachment Loss; Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: Randomised paralleled clinical trial
Who Masked: Investigator
Masking Description: All subgingival procedures were performed by the same periodontology expert, who was blinded to the placebo or AFG application.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Subgroups:control and initial pocket depths:5-6mm (Placebo Comparator): Control group divided into two subgroups according to initial pocket depths and this subgroup includes initial pocket depths:5-6mm
  Interventions: Other: placebo application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis
- Subgroups:control and initial pocket depths≥7mm (Placebo Comparator): Control group divided into two subgroups according to initial pocket depths and this subgroup includes initial pocket depths higher than 7mm
  Interventions: Other: placebo application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis
- Subgroups:AFG and initial pocket depths:5-6mm (Experimental): AFG group divided into two subgroups according to initial pocket depths and this subgroup includes initial pocket depths:5-6mm
  Interventions: Biological: autologous fibrin glue application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis
- Subgroups:AFG and initial pocket depths≥7mm (Experimental): AFG group divided into two subgroups according to initial pocket depths and this subgroup includes initial pocket depths higher than 7mm
  Interventions: Biological: autologous fibrin glue application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis

INTERVENTIONS:
Biological: autologous fibrin glue application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis — The purpose of this study was to investigate effects of autologous fibrin glue (AFG) which was an injectable platelet concentration, on clinical parameters in the nonsurgical treatment of chronic periodontitis.Seventy-two quadrants from 18 patients included in the study and divided into 2 random split-mouth groups. Control group included 631 sites (SRP+Placebo) and AFG group included 682 sites (SRP+AFG). Both groups divided into two subgroups according to initial pocket depth (PD:5-6mm and PD≥7mm).The test group was administered AFG using a blunt dental injector in the subgingival region, as an adjunct to SRP Clinical periodontal parameters including PD, clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were collected at the 1st, 3rd, and 6th months.
  Arms: Subgroups:AFG and initial pocket depths:5-6mm; Subgroups:AFG and initial pocket depths≥7mm
Other: placebo application as an adjunct to nonsurgical periodontal treatment of chronic periodontitis — Seventy-two quadrants from 18 patients included in the study and divided into 2 random split-mouth groups. Control group included 631 sites (SRP+Placebo) and AFG group included 682 sites (SRP+AFG). Both groups divided into two subgroups according to initial pocket depth (PD:5-6mm and PD≥7mm).The control group was administered placebo as an adjunct to SRP.Clinical periodontal parameters including PD, clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were collected at the 1st, 3rd, and 6th months.
  Arms: Subgroups:control and initial pocket depths:5-6mm; Subgroups:control and initial pocket depths≥7mm

SUMMARY:
Chronic periodontitis is an inflammatory and polymicrobic disease characterized by the irreversible loss of alveolar bone and connective tissue attachment of the teeth. Chronic periodontitis is the most prevalent type of periodontitis and it is seen in the great majority of the adult population.

The main objective of periodontal treatment is to heal the inflammatory tissue, to eliminate unhealthy periodontal pockets, and to reduce the number of pathogenic bacteria. The traditional treatment of chronic periodontitis is debridement performed with hand tools and ultrasonic devices. However, in deep pockets, which are difficult to access, mechanical root surface debridement is not sufficient to remove the biofilm via root instrumentation.

The regeneration of the periodontium aims at the reconstitution of the periodontal ligament, alveolar bone, and cementum. Platelet concentrates have gained popularity in regenerative periodontal therapy due to their autologous nature. Their regenerative potential is associated with growth factors such as TGFβ-1, PDGF, EGF, IGF-I, and VEGF, stimulate cell proliferation and regulate matrix remodeling and angiogenesis. Growth factors are naturally occurring proteins that regulate cell growth and development. They also modulate cell proliferation, migration, extracellular matrix formation and other cellular functions in epithelization. In addition, some growth factors may function as cell differentiation factors. These functions of the growth factors support epithelization following surgical periodontal treatment and reduce postoperative pain and swelling with their anti-inflammatory properties. Furthermore, studies have reported their antibacterial potentials.

Different platelet concentrates such as platelet-rich plasma (PRP) and platelet-rich fibrin (PRF) are obtained when whole blood is centrifuged at different speeds and for different durations. When the literature is reviewed, it is seen that these platelet concentrates are frequently used in regenerative therapies in dentistry. In 2010, Sohn et al. obtained autologous fibrin glue (AFG), an injectable platelet concentrate, by centrifuging venous blood for two minutes in a special centrifuge device (Medifuge, Silfradent, Italy; 2400-2700 rpm). AFG is used, by mixing it with bone grafts, in the production of sticky bone, which could be an alternative to titanium mesh and bone block procedures that enable grafts to remain more stable in defects.

It was found in the literature review that studies on AFG, which is a second-generation platelet concentrate, are limited in number. It was also found that these studies were conducted on sticky bone, obtained by mixing AFG with bone grafts, and there are no studies in which AFG is used alone to treat periodontal diseases. The purpose of this study is to investigate the effect of AFG, an injectable platelet concentration, on clinical parameters in the nonsurgical treatment of chronic periodontitis.

DETAILED DESCRIPTION:
This randomized controlled clinical study included patients diagnosed with moderate/severe periodontitis who applied to the Department of Periodontology, Faculty of Dentistry, Inonu University. Written consent was received from each patient. Approval was obtained from the Malatya Clinical Research Ethics Committee for our study, which was designed in compliance with the Declaration of Helsinki.

Two random split-mouth groups were formed among the patients. One side of each patient's mouth was administered AFG following SRP (test group), while the other side of the same patient's mouth was administered a placebo drug (control group).

The following periodontal parameters were evaluated in all patients before and after SRP at the 1st, 3rd, and 6th months: probing depth (PD), clinical attachment level (CAL), plaque index (PI), gingival index (GI), and bleeding on probing (BOP) index. Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 4 regions (mesiobuccal, midbuccal, distobuccal, midlingual) for PI and GI and in 6 regions (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) for PD, CAL, and BOP. Clinical attachment level was measured from the enamel-cement border. Following the initial measurement, the regions with ≥5 mm pocket depth were determined. Measurements were performed only in these regions in the 1st, 3rd, and 6th months. The initial pocket depth was considered within two subgroups as regions with 5-6 mm pocket depth and regions with ≥7 mm pocket depth.

Venous blood from each patient (9 mL) was transferred into a tube without any anticoagulant. Following the protocol recommended by Sohn et al., the venous blood collected in the tube was centrifuged in a special centrifuge machine (Medifuge, Silfradent, Italy). The AFG at the top of the tube was collected using an injector.

Nonsurgical periodontal treatments of the patients were completed in two sessions by a periodontology expert.

In the first session, the supragingival calculus was removed, and patients were given oral hygiene training and encouragement. In the second session, the SRP procedure was performed under local anesthesia in the regions in which there were periodontal pockets of ≥5 mm in the quadrants considered as the control and test groups. The test group was administered AFG using a blunt dental injector in the subgingival region, as an adjunct to SRP, while the control group was administered the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with moderate/severe chronic periodontitis;
* Being older than 18 years;
* Presence of at least three teeth in each quadrant with ≥5 mm probing pocket; depth and ≥3 mm clinical attachment loss;
* Being systemically healthy;
* Not smoking cigarettes.

Exclusion Criteria:

* Presence of a systemic disease (diabetes, hypertension, coagulopathy, radiotherapy, chemotherapy, etc.);
* Use of any drugs that could influence the results of the study;
* Periodontal treatment in the last six months before the study, or use of antibiotics in the last six months;
* Smoking or alcohol consumption;
* Pregnancy.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
change of pocket depths (PD) in millimeters at different time points | Pocket depths were evaluated in all patients at baseline and after SRP at the 1st, 3rd, and 6th months
  Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 6 regions (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) for PD.
change of clinical attachment levels (CAL) in millimeters at different time points | clinical attachment levels were evaluated in all patients at baseline and after SRP at the 1st, 3rd, and 6th months
  Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 6 regions (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) for CAL.

SECONDARY OUTCOMES:
change of bleeding on probing(BOP) scores in % at different time points | bleeding on probing scores were evaluated in all patients at baseline and after SRP at the 1st, 3rd, and 6th months
  Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 6 regions (mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, distolingual) for BOP.
change of gingival index(GI) scores in levels at different time points | gingival index scores were evaluated in all patients at baseline and after SRP at the 1st, 3rd, and 6th months
  Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 4 regions (mesiobuccal, midbuccal, distobuccal, midlingual) for GI
change of plaque index(PI) scores in levels at different time points | plaque index scores were evaluated in all patients bt baseline and after SRP at the 1st, 3rd, and 6th months
  Measurements were performed using a Williams probe (Hu-Friedy, Chicago, IL, USA) for all teeth except for the third molars, in 4 regions (mesiobuccal, midbuccal, distobuccal, midlingual) for PI.

CONTACTS AND LOCATIONS:
Overall Officials: MUSTAFA Ö USLU, Asst. Prof., Study Director — Dr.
Locations (1):
- Faculty of Dentistry, Department of Periodontology, İnonu University, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available. The outcomes of the treatment will publish in a journal and doesn't need a patient's data collection

REFERENCES:
- [Background] Heitz-Mayfield LJ, Trombelli L, Heitz F, Needleman I, Moles D. A systematic review of the effect of surgical debridement vs non-surgical debridement for the treatment of chronic periodontitis. J Clin Periodontol. 2002;29 Suppl 3:92-102; discussion 160-2. doi: 10.1034/j.1600-051x.29.s3.5.x. PMID 12787211
- [Background] The potential role of growth and differentiation factors in periodontal regeneration. J Periodontol. 1996 May;67(5):545-53. PMID 8724716
- [Background] Abdul Ameer LA, Raheem ZJ, Abdulrazaq SS, Ali BG, Nasser MM, Khairi AWA. The anti-inflammatory effect of the platelet-rich plasma in the periodontal pocket. Eur J Dent. 2018 Oct-Dec;12(4):528-531. doi: 10.4103/ejd.ejd_49_18. PMID 30369798
- [Background] Kao RT, Murakami S, Beirne OR. The use of biologic mediators and tissue engineering in dentistry. Periodontol 2000. 2009;50:127-53. doi: 10.1111/j.1600-0757.2008.00287.x. No abstract available. PMID 19388957
- [Background] Nevins M, Giannobile WV, McGuire MK, Kao RT, Mellonig JT, Hinrichs JE, McAllister BS, Murphy KS, McClain PK, Nevins ML, Paquette DW, Han TJ, Reddy MS, Lavin PT, Genco RJ, Lynch SE. Platelet-derived growth factor stimulates bone fill and rate of attachment level gain: results of a large multicenter randomized controlled trial. J Periodontol. 2005 Dec;76(12):2205-15. doi: 10.1902/jop.2005.76.12.2205. PMID 16332231
- See also: 20. Sohn D Lecture titled with sinus and ridge augmentation with CGF and AFG. In: Symposium on CGF and AFG. Tokyo, 2010. — https://www.academia.edu/22262758/Utilization_of_Autologous_Concentrated_Growth_Factors_CGF_Enriched_Bone_Graft_Matrix_Sticky_Bone_and_CGF-Enriched_Fibrin_Membrane_in_Implant_Dentistry
- See also: 21. Sohn D-S, Huang B, Kim J, Park WE,Park CC (2015) Utilization of autologous concentrated growth factors (CGF) enriched bone graft matrix (Sticky bone) and CGF-enriched fibrin membrane in Implant Dentistry. Jr Implant Adv Cli Dent 7:11-29. — https://www.academia.edu/22262758/Utilization_of_Autologous_Concentrated_Growth_Factors_CGF_Enriched_Bone_Graft_Matrix_Sticky_Bone_and_CGF-Enriched_Fibrin_Membrane_in_Implant_Dentistry